CLINICAL TRIAL: NCT06170788
Title: A Randomized, Open-label, Phase 3 Study of MK-2870 in Combination With Pembrolizumab Compared to Pembrolizumab Monotherapy in the First-line Treatment of Participants With Metastatic Non-small Cell Lung Cancer With PD-L1 TPS Greater Than or Equal to 50% (TroFuse-007)
Brief Title: Sacituzumab Tirumotecan (MK-2870) in Combination With Pembrolizumab Versus Pembrolizumab Alone in Metastatic Non-small Cell Lung Cancer (NSCLC) With Programmed Cell Death Ligand 1 (PD-L1) Tumor Proportion Score (TPS) ≥ 50% (MK-2870-007)
Acronym: TroFuse-007
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2870-007; MK-2870-007 (Other: MSD); 2023-503376-24-00 (Other: EU CT); jRCT2051240089 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); U1111-1287-1395 (Registry Identifier: UTN)
Record Dates: First submitted 2023-12-03; First posted 2023-12-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Sacituzumab tirumotecan (Experimental): Participants receive sacituzumab tirumotecan via intravenous (IV) infusion on Days 1, 15 and 29 of each 6-week cycle + 400 mg Pembrolizumab every 6 weeks (q6w) via IV infusion on Day 1 of each 6-week cycle for 18 cycles. Additionally, participants receive diphenhydramine (or equivalent), an H2 antagonist of investigator's choice, acetaminophen (or equivalent), and dexamethasone (or equivalent) per each drug's product label prior to the first 4 infusions of sacituzumab tirumotecan. At subsequent infusions, the H2 antagonist and dexamethasone are optional, at the discretion of the investigator.
  Interventions: Biological: Sacituzumab tirumotecan; Biological: Pembrolizumab; Drug: Supportive care measures
- Pembrolizumab (Active Comparator): Participants receive 400 mg Pembrolizumab via IV infusion q6w on Day 1 of each 6-week cycle for 18 cycles
  Interventions: Biological: Pembrolizumab; Drug: Supportive care measures

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — IV infusion
  Other Names: SKB264; MK-2870
  Arms: Pembrolizumab + Sacituzumab tirumotecan
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®; SCH 900475
Drug: Supportive care measures — Participants are allowed to take supportive care measures at the discretion of the investigator. Prophylactic supportive care measures may include but are not limited to antiemetic agents, antidiarrheal agents, granulocyte and erythroid growth factors, and blood transfusions

SUMMARY:
The primary objective of the study is to compare sacituzumab tirumotecan combined with pembrolizumab to pembrolizumab alone with respect to overall survival (OS). The primary hypothesis is that the combination of sacituzumab tirumotecan and pembrolizumab is superior to pembrolizumab alone with respect to OS.

All participants who have completed the first course of pembrolizumab may be eligible for up to an additional 9 cycles of pembrolizumab monotherapy if there is blinded independent central review (BICR)-verified progressive disease by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) after initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of squamous or nonsquamous NSCLC

  * Confirmation that epidermal growth factor receptor- (EGFR-), anaplastic lymphoma kinase- (ALK-), or proto-oncogene tyrosine-protein kinase ROS (ROS1-) directed therapy is not indicated as primary therapy
  * Provided tumor tissue that demonstrates programmed cell death ligand 1 (PD-L1) expression in ≥50% of tumor cells as assessed by an immunohistochemistry (IHC) central laboratory
  * An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 7 days before randomization.
  * A life expectancy of at least 3 months.
  * Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)

Exclusion Criteria:

* Diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements.
* Has Grade ≥2 peripheral neuropathy.
* History of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing.
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous clear history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea).
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease within the 6 months preceding study intervention.
* Received prior systemic anticancer therapy for their metastatic NSCLC.
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor Note: Prior treatment with an anti-PD-1, anti-PD- L1, or anti-PD-L2 agent in the neoadjuvant or adjuvant setting for nonmetastatic resectable NSCLC is allowed as long as therapy was completed at least 12 months before diagnosis of metastatic NSCLC.
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization.
* Received radiation therapy to the lung that is >30 Gy within 6 months of start of study intervention.
* Received prior radiotherapy within 2 weeks of start of study intervention, or radiation-related toxicities, requiring corticosteroids.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Known intolerance to sacituzumab tirumotecan or pembrolizumab and/or any of their excipients; for pembrolizumab, severe hypersensitivity (≥Grade 3) is exclusionary.
* Known hypersensitivity to sacituzumab tirumotecan or other biologic therapy.
* Active autoimmune disease that has required systemic treatment in the past 2 years.
* History of (noninfectious) pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD.
* Active infection requiring systemic therapy
* Concurrent active Hepatitis B and Hepatitis C virus infection.
* Human immunodeficiency virus (HIV)-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* History of allogeneic tissue/solid organ transplant.
* Requires treatment with a strong inhibitor or inducer of Cytochrome P450 3A4 (CYP3A4) at least 14 days before the first dose of study intervention and throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2028-01-25 (Estimated); Study Completion 2030-05-27 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 49 months
  OS is defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to approximately 77 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR or death due to any cause, whichever occurs first
Objective Response (OR) | Up to approximately 77 months
  The OR is defined as a confirmed complete response (CR) or partial response (PR) per RECIST 1.1 as assessed by BICR.
Duration of Response (DOR) | Up to approximately 77 months
  For participants who demonstrate confirmed CR or PR per RECIST 1.1 as assessed by BICR, duration of response is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Change from Baseline in Global Health Status/Quality of Life (QOL) [European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30) 29 Items and 30] Score | Baseline and up to approximately 77 months
  Change from baseline in the score of EORTC QLQ-C30 Items 29 and 30 will be presented. The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to Items 29 and 30 ("How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome.
Change From Baseline in Dyspnea (EORTC QLQ-C30 Item 8) Score | Baseline and up to approximately 77 months
  Change from baseline in the score of EORTC QLQ-C30 Item 8 will be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of dyspnea.
Change From Baseline in Cough (EORTC QLQ-LC13 Item 31) Score | Baseline and up to approximately 77 months
  Change from baseline in the score of EORTC QLQ-C13 Item 31 will be presented. The EORTC QLQ-C13 is a lung cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates more frequent coughing.
Change From Baseline in Chest Pain (EORTC QLQ-LC13 item 40) Score | Baseline and up to approximately 77 months
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in chest pain (EORTC QLQ-LC13 Item 40) score will be presented. A lower score indicates a better outcome.
Time to Deterioration (TTD) Based on Change From Baseline in Global Health Status (GHS)/ QOL Score (EORTC QLQ-C30 Item 29 and 30) | Up to approximately 77 months
  The TTD in GHS/QOL score (EORTC QLQ-C30 Items 29 and 30) will be presented. Participant responses to Items 29 and 30 ("How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome. TTD as assessed based on a negative change (decrease in score) from Baseline in GHS/QOL score. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) Based on Change From Baseline in Dyspnea Score (EORTC QLQ-C30 Item 8) | Up to approximately 77 months
  The TTD in Dyspnea score (EORTC QLQ-C30 Item 8) will be presented. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of dyspnea. TTD is assessed based on the time to a negative change (increase in score) from baseline. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) Based on Change From Baseline in Cough Score (EORTC QLQ-LC13 Item 31). | Up to approximately 77 months
  The TTD in Cough score (EORTC QLQ-LC13 Item 31) will be presented. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates more frequent coughing. TTD is assessed based on the time to a negative change (increase in score) from baseline. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) Based on Change From Baseline in Chest Pain Score (EORTC QLQ-LC13 Item 40) | Up to approximately 77 months
  The TTD in Chest Pain score (EORTC QLQ-LC13 Item 40) will be presented. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of chest pain. TTD is assessed based on the time to a negative change (increase in score) from baseline. A longer TTD indicates a better outcome.
Percentage of Participants That Experience at Least 1 Adverse Event | Up to approximately 77 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The percentage of participants who experience an AE will be presented.
Percentage of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 77 months
  The percentage of participants who discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (215):
- United States (15):
  - Mayo Clinic in Arizona - Phoenix ( Site 0147), Phoenix, Arizona
  - Roy and Patricia Disney Family Cancer Center - Providence Saint Joseph Medical Center ( Site 0130), Burbank, California
  - Cancer Centers of Colorado St. Mary's Regional Hospital ( Site 0132), Grand Junction, Colorado
  - Mayo Clinic in Florida-Mayo Clinic Comprehensive Cancer Center ( Site 0133), Jacksonville, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 0106), Marietta, Georgia
  - The University of Louisville, James Graham Brown Cancer Center ( Site 0121), Louisville, Kentucky
  - New England Cancer Specialists ( Site 0143), Westbrook, Maine
  - University of Massachusetts Chan Medical School-Division of Hematology/Oncology ( Site 0144), Worcester, Massachusetts
  - Allina Health Cancer Institute - Abbott Northwestern Hospital ( Site 0115), Minneapolis, Minnesota
  - Mayo Clinic - Rochester ( Site 0148), Rochester, Minnesota
  - Hattiesburg Clinic Hematology/Oncology ( Site 0104), Hattiesburg, Mississippi
  - Renown Regional Medical Center-Renown Health Medical Oncology ( Site 0134), Reno, Nevada
  - University Hospitals Cleveland Medical Center ( Site 0119), Cleveland, Ohio
  - Good Samaritan Regional Medical Center-Samaritan Pastega Regional Cancer Center ( Site 0117), Corvallis, Oregon
  - Oncology Consultants P.A. ( Site 0129), Houston, Texas
- Argentina (5):
  - Instituto Alexander Fleming ( Site 0306), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Británico de Buenos Aires-Oncology ( Site 0304), Buenos Aires, Buenos Aires F.D.
  - Centro Privado de RMI Río Cuarto S.A. II ( Site 0310), Río Cuarto, Córdoba Province
  - Instituto de Oncología de Rosario ( Site 0301), Rosario, Santa Fe Province
  - Hospital Aleman-Oncology ( Site 0300), Buenos Aires
- Australia (4):
  - Port Macquarie - Mid North Coast Cancer Institute-Medical Oncology ( Site 3002), Port Macquarie, New South Wales
  - Westmead Hospital ( Site 3000), Westmead, New South Wales
  - Grampians Health-Medical Oncology ( Site 3001), Ballarat Central, Victoria
  - Northern Hospital ( Site 3003), Epping, Victoria
- Brazil (6):
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre ( Site 0409), Porto Alegre, Rio Grande do Sul
  - Clinica Viver ( Site 0400), Santa Maria, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 0402), Barretos, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 0406), São José do Rio Preto, São Paulo
  - Instituto Nacional de Câncer - INCA ( Site 0405), Rio de Janeiro
  - Núcleo de Pesquisa Clínica da Rede São Camilo ( Site 0401), São Paulo
- Canada (3):
  - William Osler Health System ( Site 0203), Brampton, Ontario
  - Trillium Health Partners - Credit Valley Hospital ( Site 0202), Mississauga, Ontario
  - McGill University Health Centre ( Site 0200), Montreal, Quebec
- Chile (5):
  - Clinica Universidad Catolica del Maule-Oncology ( Site 0501), Talca, Maule Region
  - Orlandi Oncologia-Oncology ( Site 0504), Santiago, Region M. de Santiago
  - FALP-UIDO ( Site 0509), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0507), Santiago, Region M. de Santiago
  - Bradford Hill Norte ( Site 0516), Antofagasta
- China (32):
  - Second Affiliated hospital of Anhui Medical University ( Site 3133), Hefei, Anhui
  - Beijing Cancer hospital-intrathoratic deparmtment II ( Site 3101), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-pneumology department ( Site 3100), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital ( Site 3131), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University-Breast Surgery ( Site 3107), Xiamen, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 3134), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital-Depatrment of Respiratory and Critical Care Medicine ( Site 3108), Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University ( Site 3123), Zhanjiang, Guangdong
  - The Second Hospital of Hebei Medical University ( Site 3135), Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital-oncology of department ( Site 3132), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 3116), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 3117), Wuhan, Hubei
  - Wuhan Union Hospital ( Site 3130), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 3106), Wuhan, Hubei
  - Xiangyang Central Hospital-oncology department ( Site 3136), Xiangyang, Hubei
  - The Second Xiangya Hospital of Central South University ( Site 3138), Changsha, Hunan
  - Affiliated Hospital of Jiangnan University(Wuxi Fourth People's Hospital ) ( Site 3113), Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College ( Site 3112), Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University-Respiratory Medicine Department ( Site 3127), Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University-Oncology Department ( Site 3121), Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital ( Site 3143), Nanchang, Jiangxi
  - Jilin Province Tumor Hospital-oncology department ( Site 3126), Changchun, Jilin
  - Jinan Central Hospital-oncology department ( Site 3122), Jinan, Shandong
  - Shandong Cancer Hospital ( Site 3119), Jinan, Shandong
  - Shanghai Changhai Hospital ( Site 3125), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University ( Site 3124), Chengdu, Sichuan
  - Sichuan Cancer hospital. ( Site 3105), Chengdu, Sichuan
  - The Second People's Hospital of Neijiang ( Site 3140), Neijiang, Sichuan
  - Yunnan Province Cancer Hospital ( Site 3139), Kunming, Yunnan
  - The first Affiliated Hospital, Zhejiang University School of Medicine ( Site 3115), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine ( Site 3111), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province-Respiratory ( Site 3114), Taizhou, Zhejiang
- Colombia (3):
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0600), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 0602), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 0603), Pereira, Risaralda Department
- Czechia (4):
  - Nemocnice AGEL Ostrava - Vitkovice a.s.-Plicni oddeleni ( Site 1103), Ostrava, Ostrava Mesto
  - Multiscan-Onkologicke a radiologicke centrum Multiscan Pardubice ( Site 1105), Pardubice, Pardubický kraj
  - Vseobecna fakultni nemocnice v Praze-Onkologicka klinika ( Site 1106), Prague, Praha 2
  - Fakultni nemocnice Olomouc-Klinika plicnich nemoci a tuberkulozy ( Site 1102), Olomouc
- Denmark (3):
  - Regionshospitalet Gødstrup-Kræftklinikken ( Site 1204), Herning, Central Jutland
  - Aalborg Universitetshospital, Syd-Department of Oncology ( Site 1201), Aalborg, North Denmark
  - Odense Universitetshospital ( Site 1200), Odense, Region Syddanmark
- France (8):
  - Hôpital Saint Joseph-ONCOLOGY ( Site 1308), Marseille, Bouches-du-Rhone
  - Institut Régional du Cancer Montpellier-Medical Oncology ( Site 1309), Montpellier, Herault
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuyt-Unité d'oncologie thoracique et cutané ( Site 1303), Limoges, Limousin
  - Centre d'Oncologie de Gentilly ( Site 1301), Nancy, Meurthe-et-Moselle
  - Centre Hospitalier de la Côte Basque ( Site 1300), Bayonne, Pyrenees-Atlantiques
  - L HOPITAL NORD OUEST ( Site 1310), Gleizé, Rhone
  - Clinique de l'Europe-Service de pneumologie ( Site 1304), Amiens, Somme
  - Centre Hospitalier Universitaire de Poitiers-Pôle régional de cancérologie ( Site 1305), Poitiers, Vienne
- Germany (11):
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen-Medizinische Klinik V ( Site 1409), München, Bavaria
  - Klinikum Bogenhausen-Klinik für Pneumologie und Onkologische Pneumologie ( Site 1406), München, Bavaria
  - Klinikum Nürnberg Nord-5. Med. Klinik ( Site 1407), Nuremberg, Bavaria
  - Universitätsklinikum Marburg-Comprehensive Cancer Center ( Site 1412), Marburg, Hesse
  - Medizinische Hochschule Hannover-Department of Pneumology ( Site 1411), Hanover, Lower Saxony
  - Bethanien Krankenhaus Moers ( Site 1400), Moers, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus-Medizinische Klinik A ( Site 1410), Münster, North Rhine-Westphalia
  - Universitätsmedizin Johannes Gutenberg Universität Mainz- Klinik für Pneumologie ( Site 1404), Mainz, Rhineland-Palatinate
  - LungenClinic Grosshansdorf-Onkologie ( Site 1401), Großhansdorf, Schleswig-Holstein
  - SRH Wald-Klinikum Gera-Zentrum für klinische Studien ( Site 1403), Gera, Thuringia
  - Charité Campus Virchow-Klinikum-Department of Infectious Diseases and Pulmonary Medicine ( Site 1402), Berlin
- Italy (7):
  - Instituto Tumori Giovanni Paolo II-SSD Oncologia Medica per la Patologia Toracica ( Site 1804), Bari, Apulia
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori"-Oncologia Medica ( Site 1807), Meldola, Emilia-Romagna
  - P.O. "S. Maria della Misericordia" Azienda Sanitaria Univers-Oncology Department ( Site 1803), Udine, Friuli Venezia Giulia
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1800), Milan, Lombardy
  - AOU Renato Dulbecco ( Site 1801), Catanzaro
  - Azienda Ospedaliera Universitaria Careggi ( Site 1809), Florence
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 1806), Roma
- Japan (30):
  - Fujita Health University Hospital ( Site 3411), Toyoake, Aichi-ken
  - Hirosaki University Hospital ( Site 3429), Hirosaki, Aomori
  - National Cancer Center Hospital East ( Site 3403), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 3415), Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center ( Site 3417), Fukuoka, Fukuoka
  - Kurume University Hospital ( Site 3418), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 3402), Ōta, Gunma
  - National Hospital Organization Himeji Medical Center ( Site 3426), Himeji, Hyōgo
  - Iwate Medical University Hospital ( Site 3428), Shiwa-gun, Iwate
  - St. Marianna University Hospital ( Site 3421), Kawasaki, Kanagawa
  - Yokohama Municipal Citizen's Hospital ( Site 3425), Yokohama, Kanagawa
  - Kanagawa Cancer Center ( Site 3408), Yokohama, Kanagawa
  - Matsusaka Municipal Hospital ( Site 3422), Matsusaka, Mie-ken
  - Tohoku University Hospital ( Site 3424), Sendai, Miyagi
  - Sendai Kousei Hospital ( Site 3400), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 3412), Hirakata, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 3413), Takatsuki, Osaka
  - National Hospital Organization Ureshino Medical Center ( Site 3427), Ureshino, Saga-ken
  - Niigata Cancer Center Hospital ( Site 3409), Niigata, Saitama
  - Shizuoka Cancer Center ( Site 3410), Suntogun, Shizuoka
  - Dokkyo Medical University Hospital ( Site 3401), Shimotsugagun, Tochigi
  - Tokyo Metropolitan Komagome Hospital ( Site 3405), Bunkyo, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 3404), Koto, Tokyo
  - Toho University Omori Medical Center ( Site 3420), Ōta-ku, Tokyo
  - Tokyo Medical University Hospital ( Site 3407), Shinjuku, Tokyo
  - National Center for Global Health and Medicine ( Site 3406), Shinjuku, Tokyo
  - National Hospital Organization Yamaguchi Ube Medical Center ( Site 3423), Ube, Yamaguchi
  - National Hospital Organization Kyushu Medical Center ( Site 3416), Fukuoka
  - Saiseikai Kumamoto Hospital ( Site 3419), Kumamoto
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 3414), Osaka
- Mexico (6):
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 0715), Guadalajara, Jalisco
  - Higiea Oncologia ( Site 0721), Mexico City, Mexico City
  - Axis Heilsa S. de R.L. de C.V. ( Site 0719), Monterrey, Nuevo León
  - Centro de Atención e Investigación Cardiovascular del Potosí ( Site 0713), San Luis Potosí City, San Luis Potosí
  - Oaxaca Site Management Organization S.C. ( Site 0718), Oaxaca City
  - Clinica Integral Internacional de Oncología ( Site 0714), Puebla City
- Netherlands (3):
  - Amphia Ziekenhuis, locatie Breda Molengracht-long oncologie ( Site 1901), Breda, North Brabant
  - ETZ Elisabeth-Department of Pulmonary Diseases ( Site 1902), Tilburg, North Brabant
  - Isala, locatie Zwolle-Poli Longziekten ( Site 1903), Zwolle, Overijssel
- Peru (5):
  - Clinica Vallesur - AUNA ( Site 0854), Arequipa, Ariqipa
  - Detecta Clínica ( Site 0853), Surquillo, Muni Metro de Lima
  - IPOR Instituto Peruano de Oncología & Radioterapia-Centro de Investigación ( Site 0851), Lima
  - INSTITUTO NACIONAL DE ENFERMEDADES NEOPLASICAS ( Site 0850), Lima
  - Hospital Cayetano Heredia-Oncology ( Site 0855), Lima
- Poland (8):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 2003), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Regionalny Szpital Specjalistyczny im. dr. Władyslawa Biegańskiego ( Site 2013), Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Wojewodzki Szpital Zespolony im Ludwika Rydygiera w Toruniu ( Site 2016), Torun, Kuyavian-Pomeranian Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie-Oncology Department ( Site 2015), Krakow, Lesser Poland Voivodeship
  - Instytut Gruźlicy i Chorób Płuc w Warszawie-3rd Dep of Lung Diseases and Oncology ( Site 2011), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 2000), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 2001), Przemyśl, Podkarpackie Voivodeship
  - SPZOZ Uniwersytecki Szpital Kliniczny Im. Wojskowej Akademii Medycznej UM W Łodzi Centralny Szpital ( Site 2012), Lodz, Łódź Voivodeship
- Portugal (5):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil ( Site 2104), Lisbon, Lisbon District
  - Unidade Local de Saude de Santa Maria - Hospital Pulido Valente ( Site 2101), Lisbon, Lisbon District
  - Hospital Dr. Nélio Mendonça ( Site 2105), Funchal, Madeira
  - Unidade Local de Saude Gaia/Espinho - Hospital Eduardo Santos Silva ( Site 2103), Vila Nova de Gaia, Porto District
  - Hospital CUF - Tejo ( Site 2100), Lisbon
- South Korea (8):
  - Wonju Severance Christian Hospital ( Site 3808), Wŏnju, Kang-won-do
  - National Cancer Center ( Site 3801), Goyang-si, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital-Medical Oncology ( Site 3800), Suwon, Kyonggi-do
  - Ajou University Hospital-Hematology-Oncology ( Site 3806), Suwon, Kyonggi-do
  - Chungbuk National University Hospital-Internal medicine ( Site 3804), Cheongju-si, North Chungcheong
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 3807), Daegu, Taegu-Kwangyokshi
  - Asan Medical Center-Lung Cancer Center ( Site 3805), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 3802), Seoul
- Spain (8):
  - Hospital Jerez de la Frontera-UGC Oncología ( Site 2333), Jerez de la Frontera, Cadiz
  - CHUAC-Hospital Teresa Herrera-MEDICAL ONCOLOGY ( Site 2335), A Coruña, La Coruna
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 2331), Pozuelo de Alarcón, Madrid
  - H.R.U Malaga - Hospital General ( Site 2332), Málaga, Malaga
  - Fundación Instituto Valenciano de Oncología-Oncologico ( Site 2336), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 2330), Barcelona
  - Hospital La Princesa ( Site 2338), Madrid
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Medical Oncology ( Site 2337), Seville
- Taiwan (11):
  - Chi Mei Hospital - Liouying Branch ( Site 3908), Tainan, Tainan
  - National Taiwan University Cancer Center (NTUCC) ( Site 3907), Taipei City, Taipei
  - National Taiwan University Hospital - Hsinchu branch ( Site 3901), Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 3904), Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 3902), Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital ( Site 3912), New Taipei City
  - Taichung Veterans General Hospital-Chest ( Site 3905), Taichung
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 3903), Tainan
  - Chi Mei Medical Center ( Site 3915), Tainan
  - National Taiwan University Hospital-Oncology ( Site 3906), Taipei
  - Mackay Memorial Hospital ( Site 3909), Taipei
- Thailand (3):
  - Chulalongkorn University-Medicine ( Site 4003), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 4000), Bangkok, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital-Chiang Mai Clinical Trial Unit (CM-CTU) ( Site 4001), Chiang Mai
- Turkey (Türkiye) (11):
  - Medipol Mega Universite Hastanesi-oncology ( Site 2508), Stanbul, Istanbul
  - Ege Universitesi Hastanesi-Chest Diseases Department ( Site 2503), Bornova, İzmir
  - Erciyes University ( Site 2511), Talas, Kayseri
  - Adana Medical Park Seyhan Hastanesi-Medikal Onkoloji ( Site 2507), Adana
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi-oncology ( Site 2506), Ankara
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 2501), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 2505), Ankara
  - Ankara Bilkent Şehir Hastanesi ( Site 2500), Ankara
  - Pamukkale University Medical Faculty, Fahri Goksin Oncology Centre-Oncolgyy-Hematology ( Site 2510), Denizli
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 2502), Istanbul
  - Ondokuz Mayıs Universitesi ( Site 2509), Samsun
- United Kingdom (5):
  - Royal Free Hospital ( Site 2601), London, England
  - Queen Alexandra Hospital-Oncology Department ( Site 2603), Portsmouth, Hampshire
  - Kent and Canterbury Hospital-Oncology Research ( Site 2606), Canterbury, Kent
  - Guy's & St Thomas' NHS Foundation Trust-Oncology & Haematology Clinical Trials ( Site 2605), London, London, City of
  - James Cook University Hospital ( Site 2604), Central Middlesbrough, Middlesbrough
- Vietnam (6):
  - National Lung Hospital-Oncology Department ( Site 4175), Hanoi, Hanoi
  - Tam Anh General Hospital ( Site 4179), Hanoi, Hanoi
  - Cho Ray Hospital ( Site 4171), Ho Chi Minh, Hanoi
  - K Hospital - National Cancer Hospital ( Site 4174), Hà Nội
  - Ho Chi Minh City Oncology Hospital - Tan Phu Ward ( Site 4173), Ho Chi Minh City
  - Thong Nhat Hospital ( Site 4170), Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26171&tenant=MT_MSD_9011